CLINICAL TRIAL: NCT02650934
Title: Predictors of Heart Failure After ST-segment Elevation Myocardial Infarction (HF-EXPRESS)
Acronym: HF-EXPRESS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Nafiz Korez Sincan State Hospital (Other Government)
Collaborators: Ankara Diskapi Training and Research Hospital (Other); Ankara City Hospital Bilkent (Other); Ankara Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 114S309
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-06

CONDITIONS: Heart Failure and ST Elevation Myocardial Infarction
Keywords: STEMI, Heart Failure, Inflammation, Haptoglobin Polymorphisms, Adverse Remodeling, Genetics, GWAS, MRI
MeSH Terms: conditions — Heart Failure; ST Elevation Myocardial Infarction; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood specimen
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Adverse remodelling: EF below 40% following MI and remain below 40% after reperfusion
  Interventions: Procedure: Percutanous coronary intervention
- not adverse remodelling: EF below 40% following MI and remodelling after reperfusion or EF above 40 % following MI
  Interventions: Procedure: Percutanous coronary intervention

INTERVENTIONS:
Procedure: Percutanous coronary intervention

SUMMARY:
Objective: The purpose of this project is to study the post miyocardial infaction (MI) damage and subsequently developed post-infarct cardiac repair process on the basis of cellular, molecular and imaging techniques. Besides this, whole genomesequencing and analysis (GWAS) will be performed to determine common varying genetic loci in order to anticipate whetherthese findings and its related pathways would be the predictors of adverse remodeling after MI or not.

DETAILED DESCRIPTION:
A brief description of the issue and the original value of the subject: Epidemiological studies show a clear increase ininfarct-related complications due to increased survival after MI and aging population. Heart failure is the most prevalent complication after MI, which has reached epidemic proportions in western societies. For the period between 2010 and 2030,according to projections made in developed countries, about 10% increment in all cardiovascular disease is being predictedhowever increment in heart failure (HF) would be such a dramatic figure which is about 25%. HF is an increasing burden tosociety and healthcare systems, since its prevalence and incidence is dramatically increasing. There has not been aprospective study that assesses the exact cellular and geometric course after MI in human. This study will allow us tounderstand the behavior of cells involved in cardiac repair after MI. In addition, it will show us the exact functional andgeometric course after MI. Finally, the current study will also provide novel diagnostic and therapeutic targets via genomic andproteomic studies. All together, we envision to find new efficient ways to identify/treat patients at risk to develop HF after MI.

ELIGIBILITY:
Inclusion Criteria:

18-80 years old patients with myocardial infarction in the first 12 hours TIMI 3 flow following PCI

Exclusion Criteria:

Right ventiricular myocardial infarction Cardiogenic shock History of CABG, PCI or valvular disease History of Cardiomyopathy severe LV hypertrophy No reflow after PCI Chronic kidney disease (GFR<60) Systemic inflammatory disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-80 years old patients with myocardial infarction in the first 12 hours
Sampling Method: Probability Sample
Enrollment: 312 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular death, nonfatal MI, stroke | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Omer Sahin, MD, Study Chair — Dr.Nafiz Korez state hospital
Locations (1):
- Dr.Nafiz Korez state hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Orn S, Ueland T, Manhenke C, Sandanger O, Godang K, Yndestad A, Mollnes TE, Dickstein K, Aukrust P. Increased interleukin-1beta levels are associated with left ventricular hypertrophy and remodelling following acute ST segment elevation myocardial infarction treated by primary percutaneous coronary intervention. J Intern Med. 2012 Sep;272(3):267-76. doi: 10.1111/j.1365-2796.2012.02517.x. Epub 2012 Feb 26. PMID 22243053
- [Result] Palazzuoli A, Beltrami M, Gennari L, Dastidar AG, Nuti R, McAlindon E, Angelini GD, Bucciarelli-Ducci C. The impact of infarct size on regional and global left ventricular systolic function: a cardiac magnetic resonance imaging study. Int J Cardiovasc Imaging. 2015 Jun;31(5):1037-44. doi: 10.1007/s10554-015-0657-3. Epub 2015 Apr 12. PMID 25863669
- [Result] Scott AE, Semple SI, Redpath TW, Hillis GS. Low-dose dobutamine adds incremental value to late gadolinium enhancement cardiac magnetic resonance in the prediction of adverse remodelling following acute myocardial infarction. Eur Heart J Cardiovasc Imaging. 2013 Sep;14(9):906-13. doi: 10.1093/ehjci/jes320. Epub 2013 Jan 12. PMID 23313958